CLINICAL TRIAL: NCT01352325
Title: Randomized Controlled Trial on the Efficacy of System Constellations on Psychological Well-being in a General Population Based Sample
Brief Title: Efficacy of System Constellations in a General Population
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Jochen Schweitzer-Rothers, Professor, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFBC11; SFB 619 project C11 (Other: German Research Council)
Record Dates: First submitted 2011-05-04; First posted 2011-05-11 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Psychological Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- system constellations seminar (exp. group) (Experimental): Study participants randomized to this group receive the intervention (system constellation seminar) 4 months prior to the control group
  Interventions: Behavioral: system constellations seminar
- system constellations seminar (control group) (Experimental): Study participants randomized to this group receive the intervention (system constellations seminar) 4 months after the experimental group.
  Interventions: Behavioral: system constellations seminar

INTERVENTIONS:
Behavioral: system constellations seminar — individual-centered intervention in a group setting, duration 3 days
  Arms: system constellations seminar (exp. group)
Behavioral: system constellations seminar — individual-centered intervention in a group setting, duration 3 days
  Arms: system constellations seminar (control group)

SUMMARY:
The purpose of this study is to investigate the efficacy of system constellations in a monocentric, single-masked randomized controlled trial.

The method of system constellations refers to an approach which integrates ideas from family systems therapy with elements from psychodrama. The constellations are conducted in a group based seminar-setting, each seminar lasting three days.

Based on the model of a general psychotherapy and the consistency theory, the effects of system constellations on psychological functioning are explored.

It is predicted that participation in a system constellation seminar changes the level of psychological functioning at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* agreement to participate in a 3-day system constellations seminar
* agreement to be randomized into treatment group or control group (waiting condition)
* agreement not to participate in another system constellation seminar until completion of study

Exclusion Criteria:

* acute suicidal tendency
* acute psychotic episode
* acute drug or alcohol intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in psychological well-being at 2 weeks and four months | Baseline, day of treatment, 2 weeks after treatment, 4 months after treatment
  Psychological well-being will be assessed using the 'Outcome Questionnaire' in its German version (EB-45). The EB-45 is a brief 45-item self report outcome/tracking instrument designed for repeated measurement of client progress through the course of psychotherapy and following termination. The scales of the EB-45 measure symptom distress, interpersonal functioning, and social role.

SECONDARY OUTCOMES:
Change from Baseline in Psychological distress after 2 weeks and 4 months | Baseline, day of treatment, 2 weeks after treatment, 4 months after treatment
  The FEP-2, 40-item self report questionnaire, measures psychological distress according to the phase model of therapeutic change as well as the interpersonal model of psychological distress.
Change from Baseline in Incongruence at 2 weeks and 4 months | Baseline, day of treatment, 2 weeks after treatment, 4 months after treatment
  Motivational incongruence is defined as the unsatisfactory realization of motivational goals and is based on the concept of General Psychotherapy by Klaus Grawe. The Incongruence Questionnaire (INK) is an instrument that assesses motivational incongruence, defined as the discrepancy between a person's motivational goals and his/her perception of reality. The short version of this questionnaire that will be used in our study (K-INK) comprises 23 items.
Goal achievement at 2 weeks and 4 months | day of treatment, 2 weeks after treatment, 4 months after treatment
  Goal achievement will be assessed using Goal Attainment Scaling as a method for the assimilation of achievement in a number of individually set goals into a single aggregated 'goal attainment score', providing a person-centred outcome, focused on that individual's priorities. Goal attainment scaling is operationalized by an open-ended question, in which study participants descriobe their individual goals. In a second step these goals will be coded according to the Bern inventory of psychotherapy goals (BIT-C).
Change from Baseline in 'Experiences in family and organisational systems' at 2 weeks and 4 months | day of treatment, 2 weeks after treatment, 4 months after treatment
  The subjective quality of family and organizational systems will be assessed by the HFES (Heidelberger Fragebogen zum Erleben in Systemen: Heidelberg Questionnaire on experiences in systems), a self-constructed questionnaire comprising 24 items.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Schweitzer-Rothers, Professor, Study Director — Institute of Medical Psychology, University Hospital Heidelberg/Germany
Locations (1):
- Institute of Medical Psychology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Hunger C, Bornhauser A, Link L, Schweitzer J, Weinhold J. Improving experience in personal social systems through family constellation seminars: results of a randomized controlled trial. Fam Process. 2014 Jun;53(2):288-306. doi: 10.1111/famp.12051. Epub 2013 Nov 19. PMID 24251855